CLINICAL TRIAL: NCT02780869
Title: Prospective, Randomized, Controlled, Multicenter, Pivotal, Clinical Investigation Evaluating the Safety and Efficacy of HEMOBLAST Bellows in Cardiothoracic, Abdominal, and Orthopedic Lower Extremity Surgeries
Brief Title: HEMOBLAST Pivotal Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETC 2015-002
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Hemostasis
MeSH Terms: interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational (Experimental): HEMOBLAST Bellows
  Interventions: Device: HEMOBLAST Bellows
- Control (Active Comparator): Absorbable gelatin sponge, USP with thrombin
  Interventions: Device: Absorbable gelatin sponge, USP with thrombin

INTERVENTIONS:
Device: HEMOBLAST Bellows
  Arms: Investigational
Device: Absorbable gelatin sponge, USP with thrombin
  Arms: Control

SUMMARY:
The purpose of this prospective, randomized, controlled study is to evaluate the safety and efficacy of a new hemostatic device (HEMOBLAST™ Bellows) compared to a control device, absorbable gelatin sponge USP with thrombin.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is undergoing an elective open cardiothoracic, abdominal, or orthopedic lower extremity surgery;

  * Subject or an authorized legal representative is willing and able to give prior written informed consent for investigation participation;
  * Subject undergoing cardiothoracic surgery is not allergic to protamine; and
  * Subject is 21 years of age or older.

Exclusion Criteria:

* • Subject is undergoing a laparoscopic, thoracoscopic, or robotic surgical procedure;

  * Subject is undergoing a neurologic surgical procedure;
  * Subject is undergoing a spinal surgical procedure;
  * Subject is undergoing an emergency surgical procedure;
  * Subject is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding;
  * Subject has a clinically significant coagulation disorder or disease, defined as a platelet count < 100,000 per microliter or International Normalized Ratio > 1.5 within 4 weeks of surgery;
  * Subject receiving intravenous heparin within 12 hours before surgery or oral Coumadin within 2 days before surgery;
  * Subject receiving antiplatelet medications within 5 days prior to surgery;
  * Subject undergoing abdominal or orthopedic lower extremity surgery receiving aspirin within 7 days prior to surgery;
  * Subject has an active or suspected infection at the surgical site;
  * Subject has had or has planned to receive any organ transplantation;
  * Subject has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
  * Subject has ASA classification of 5;
  * Subject has a life expectancy of less than 3 months;
  * Subject has a known psychiatric disorder, which in the opinion of the Principal Investigator, would preclude the subject from completing this clinical study;
  * Subject has a documented severe congenital or acquired immunodeficiency;
  * Subject has religious or other objections to porcine, bovine, or human components;
  * Subject in whom the investigational or control device will be used at the site of a valve replacement or repair;
  * Subject in whom the investigational or control device will be used at the site of a synthetic graft or patch implant;
  * Subject is currently participating or has participated in another clinical trial within the past 30 days and is receiving/has received an investigational drug, device, or biologic agent; and
  * Subject is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator.

Intraoperative Eligibility Criteria:

* Subject does not have an active or suspected infection at the surgical site;
* Subject undergoing cardiothoracic surgery with anticoagulation must have anticoagulation reversed prior to target bleeding site (TBS) identification and treatment;
* Subject in whom the Investigator is able to identify a TBS for which any applicable conventional means for hemostasis are ineffective or impractical; and
* Subject has a TBS with an SBSS score of 1, 2, or 3.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Chapman, MD, Principal Investigator — Washington University School of Medicine
Locations (17):
- United States (17):
  - CORE Institute, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Lotus Clinical Research, Pasadena, California
  - Miami Plastic Surgery, Miami, Florida
  - Queens Medical Center, Honolulu, Hawaii
  - Suburban Hospital - Johns Hopkins Medicine, Bethesda, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Hanover, New Hampshire
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Hunstad Kortesis Center, Huntsville, North Carolina
  - Intermountain Liver Disease and Transplant Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Spectrum Medical, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject completed follow-up: August 19, 2016 Last patient completed follow-up: January 18, 2017
Pre-assignment Details: Subject enrollment occurred after the subject met preoperative eligibility criteria, gave written informed consent, and met intraoperative eligibility criteria. Subjects were randomized and treated subsequent to enrollment. Subjects could withdraw or be withdrawn from the study at any time after enrollment, including prior to treatment.
Period: Overall Study
Arm/Group | Investigational | Control
Started | 175 | 83
Completed | 162 | 74
Not Completed | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational | Control | Total
Number analyzed (Participants) | 175 | 83 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (14.79) | 56.2 (14.62) | 56.7 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 49 | 155
  Male | 69 | 34 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 7 | 24
  Not Hispanic or Latino | 157 | 76 | 233
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 6 | 3 | 9
  Black or African American | 25 | 14 | 39
  White | 123 | 57 | 180
  More than one race | 11 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Hemostasis
Description: The proportion of subjects achieving hemostasis at 6 minutes post-hemostat application was calculated. Hemostasis was defined as a grade of 0 (None/Dry) on the Surface Bleeding Severity Scale, with additional grades, ranging from 1 (Minimal/Oozing) to 5 (Extreme/Gushing), considered a failure of hemostasis.
Time Frame: Intraoperative, 6 Minutes Post-Application
Population: The efficacy analysis population was defined as the Time-To-Hemostasis (TTH) population and included all subjects who were randomized, received study intervention, and had a TTH assessment recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 159 | 83
Participants | 148 | 61
Statistical Analysis 1: Comparison: Investigational vs Control; Test type: Non-Inferiority — The primary endpoint was designed to establish comparable efficacy based upon a non-inferiority margin of 10% for the difference in the probability of TTH within 6 minutes comparing HEMOBLAST™ to G+T (HEMOBLAST™- G+T). Letting θ denote the true difference in the probability of hemostasis at 6 minutes between HEMOBLAST™ to G+T, the trial will test the null hypothesis H0: θ ≤ -0.10 vs. the alternative hypothesis HA : θ > -0.10 using a one-sided level 0.025 test; p < 0.0001, Cochran-Mantel-Haenszel; Stratified adjustments for surgery type were made using the Cochran-Mantel-Haenszel weighting
Statistical Analysis 2: Comparison: Investigational vs Control; A secondary endpoint of superiority of HEMOBLAST relative to G+T for success at achieving hemostasis within 6 minutes was evaluated; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Adjustment for mulitple comparisons were made when assessing secondary endpoints using a fixed sequence closed testing procedure to control the family-wise type I error rate at 0.05

2. Secondary Outcome: Product Preparation Time
Description: The average time from the opening of the package to the product being ready to use, measured in minutes and seconds.
Time Frame: Intraoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Investigational | Control
Number analyzed (Participants) | 159 | 83
Minutes | 0.37 (0.16) | 2.40 (0.794)
Statistical Analysis 1: Comparison: Investigational vs Control; The difference in mean preparation time was tested using a linear regression model with stratified adjustment for surgery type; Test type: Superiority; p < 0.0001, Regression, Linear — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Proportion of Subjects Achieving Hemostasis
Description: The proportion of subjects achieving hemostasis at 3 minutes post-hemostat application was calculated
Time Frame: Intraoperative, 3 Minutes Post-Application
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 159 | 83
Participants | 113 | 38
Statistical Analysis 1: Comparison: Investigational vs Control; Test type: Non-Inferiority — The difference in the probability of hemostasis within 3 minutes was tested using a logistic regression model with stratified adjustment for surgery type; p < 0.0001, Regression, Logistic — Adjustment for multiple comparisons when assessing secondary endpoints was performed using a fixed sequence closed testing procedure to control the family-wise type I error rate at 0.05
Statistical Analysis 2: Comparison: Investigational vs Control; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Enrollment until completion of 6-week follow-up visit
Description: All adverse events (AEs) through final follow-up were collected. An AE is defined according to the European Standard EN ISO 14155 as 'any untoward medical occurrence in a subject.' An AE related to a device (adverse device effect, ADE) is defined as 'any untoward and unintended response to an investigational medical device.'
Arm/Group | Investigational | Control
All-Cause Mortality (participants affected / at risk) | 0/175 | 3/83
Serious Adverse Events (participants affected / at risk) | 19/175 | 11/83
Other Adverse Events (participants affected / at risk) | 84/175 | 47/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational (N=175) | Control (N=83)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 3 | 2
Death (General disorders) | 0 | 3
Delirium (Nervous system disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Ascites (General disorders) | 1 | 0
Pleural effusion (General disorders) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hemothorax (General disorders) | 1 | 0
Hypotension (General disorders) | 0 | 2
Bacteremia (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 3 | 0
Melena (General disorders) | 0 | 1
Nausea (General disorders) | 1 | 0
Aortic dissection (Cardiac disorders) | 1 | 0
RA lead dislodgement (Product Issues) | 0 | 1 — RA lead dislodgement
Right bronchopleural fistula (Surgical and medical procedures) | 1 | 0
Pain (General disorders) | 1 | 0
Respiratory insufficiency (General disorders) | 2 | 1
Skin rash/hives (Immune system disorders) | 1 | 0
Syncope (General disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pulmonary embolism (General disorders) | 1 | 0
Stroke (General disorders) | 1 | 1
Vomiting (General disorders) | 1 | 0
Dehisence (Skin and subcutaneous tissue disorders) | 1 | 1
Seroma (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational (N=175) | Control (N=83)
Abnormal bloodwork (Blood and lymphatic system disorders) | 13 | 5
Anemia (Blood and lymphatic system disorders) | 10 | 9
Constipation/ileus (Gastrointestinal disorders) | 12 | 5
Arrythmia (Cardiac disorders) | 16 | 7
Fluid overload (General disorders) | 8 | 5
Infection (Infections and infestations) | 7 | 6 — Non wound-related
Nausea (General disorders) | 15 | 3
Pain (General disorders) | 25 | 11
Wound related (Skin and subcutaneous tissue disorders) | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT02780869/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02780869/SAP_001.pdf